CLINICAL TRIAL: NCT03784963
Title: Open-Label Prospective Randomized Control Trial to Investigate the Efficacy of Omega-3 Fatty Acid Therapy in Preventing Gastrointestinal Bleeding in Patients With Continuous-Flow Left Ventricular Assist Device
Brief Title: Efficacy of Omega-3 Fatty Acid Therapy in Preventing Gastrointestinal Bleeding in Patients With CF-LVAD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB18-0576
Record Dates: First submitted 2018-12-03; First posted 2018-12-24 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Heart Failure; Gastrointestinal Bleeding
Keywords: Angiogenesis; Inflammation; Microbiome
MeSH Terms: conditions — Heart Failure; Gastrointestinal Hemorrhage; Inflammation | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Primary Prevention Intervention (Experimental): In patients with CF-LVAD who have not had a gastrointestinal bleed, patients randomized to intervention will receive 4 grams of Nature Made Ultra Omega-3 Fish Oil once daily for 1 year along with standard of care.
  Interventions: Drug: Omega 3 fatty acids
- Primary Prevention Non-Intervention (Placebo Comparator): In patients with CF-LVAD who have not had a gastrointestinal bleed, patients randomized to placebo will receive no fish oil and only standard of care.
  Interventions: Other: Placebo
- Secondary Prevention Intervention (Experimental): In patients with CF-LVAD who have had a gastrointestinal bleed, patients randomized to intervention will receive 4 grams of Nature Made Ultra Omega-3 Fish Oil once daily for 1 year along with standard of care.
  Interventions: Drug: Omega 3 fatty acids
- Secondary Prevention Non-Intervention (Placebo Comparator): In patients with CF-LVAD who have had a gastrointestinal bleed, patients randomized to placebo will receive no fish oil and only standard of care.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Omega 3 fatty acids — Patients will receive 4 grams fish oil once daily
  Arms: Primary Prevention Intervention; Secondary Prevention Intervention
Other: Placebo — Standard of care
  Arms: Primary Prevention Non-Intervention; Secondary Prevention Non-Intervention

SUMMARY:
This study evaluates the efficacy of high-dose fish oil in decreasing rates of gastrointestinal bleeding in patients with continuous-flow left ventricular assist devices. Half of the patients without history of bleeding will receive fish oil while the other half will not. Half of the patients with history of bleeding will receive fish oil while the other half will not. Markers of angiogenesis and inflammation, as well as changes in the microbiome will be assessed in each group.

DETAILED DESCRIPTION:
A potential mechanism of bleeding in patients with continuous-flow left ventricular assist devices (CF-LVAD) is dysfunctional angiogenesis. Angiogenesis is a complicated process controlled by several markers. Previous studies have shown that elevated Angiopoietin-2 and TNF-alpha are associated with bleeding events in CF-LVAD patients.

Fish oil has anti-inflammatory and potentially anti-angiogenic properties. A retrospective study of CF-LVAD patients on high-dose fish oil showed a marked decrease in gastrointestinal bleeding rates in these patients. Additionally, these patients had lower levels of circulating Angiopoietin-2. Fish oil is known to have an effect on the microbiome, and the aforementioned effects may be seen in changes of the microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed consent
2. Age > 18 years
3. Subjects with a CF-LVAD or are scheduled to receive a CF-LVAD implant

Exclusion Criteria:

1. Psychiatric disorder or disease, irreversible cognitive dysfunction or psychosocial issues that might impair compliance with the study.
2. Patients already taking fish oil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Nguyen, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study terminated by PI for low/no enrollment prior to primary and secondary endpoints. All efforts were taken to gather all possible data.
Period: Overall Study
Arm/Group | Primary Prevention Intervention | Primary Prevention Non-Intervention | Secondary Prevention Intervention | Secondary Prevention Non-Intervention
Started | 12 | 10 | 1 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 12 | 10 | 1 | 0
Not completed — Study terminated by PI for low/no enrollment. All efforts were taken to gather all possible data. | 12 | 10 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated by PI for low/no enrollment prior to primary and secondary endpoints. All efforts were taken to gather all possible data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Prevention Intervention | Primary Prevention Non-Intervention | Secondary Prevention Intervention | Secondary Prevention Non-Intervention | Total
Number analyzed (Participants) | 12 | 10 | 1 | 0 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [49 to 59.5] | 53.5 [37 to 73] | 76 [76 to 76] |  | 55 [49 to 59.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 0 | 0 | 5
  Male | 9 | 8 | 1 | 0 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 5 | 0 | 0 | 13
  White | 4 | 5 | 0 | 0 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ischemic [Count of Participants; unit: Participants]
  Ischemic | 4 | 2 | 1 | 0 | 7
  Non-Ischemic | 8 | 8 | 0 | 0 | 16
Dilated Cardiomyopathy [Count of Participants; unit: Participants] — Dilated cardiomyopathy is etiology of heart failure and a disease of the heart muscle of the left ventricle, specifically in its ability to dilate.
  Participants
    Dilated | 7 | 8 | 0 | 0 | 15
    Not Dilated | 5 | 2 | 1 | 0 | 8
Diabetes Mellitus (DM) [Count of Participants; unit: Participants]
  Diabetes Mellitus | 7 | 2 | 1 | 0 | 10
  No Diabetes Mellitus | 5 | 8 | 0 | 0 | 13
Hypertension (HTN) [Count of Participants; unit: Participants]
  Hypertension | 7 | 5 | 1 | 0 | 13
  No Hypertension | 5 | 5 | 0 | 0 | 10
Cerebrovascular accident and Stroke (CVA) [Count of Participants; unit: Participants]
  Cerebrovascular accident and Stroke | 2 | 0 | 0 | 0 | 2
  No Cerebrovascular accident and Stroke | 10 | 10 | 1 | 0 | 21
Obstructive Sleep Apnea (OSA) [Count of Participants; unit: Participants]
  Obstructive Sleep Apnea | 5 | 2 | 0 | 0 | 7
  No Obstructive Sleep Apnea | 7 | 8 | 1 | 0 | 16
Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants]
  Chronic Obstructive Pulmonary Disease | 4 | 0 | 1 | 0 | 5
  No Chronic Obstructive Pulmonary Disease | 8 | 10 | 0 | 0 | 18
Pre-LVAD Implant New York Heart Association Class (NYHA) [Count of Participants; unit: Participants] — NYHA class determines the functional status of the patient. There are classes I-IV. Class I is no symptoms and IV is symptoms at rest.
  Participants
    1 | 0 | 0 | 0 | 0 | 0
    2 | 1 | 1 | 0 | 0 | 2
    3 | 2 | 2 | 0 | 0 | 4
    4 | 9 | 7 | 1 | 0 | 17
Interagency Registry for Mechanically Assisted Circulatory Support (Intermacs) [Count of Participants; unit: Participants] — The Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) identifies patients with advanced heart failure undergoing mechanical circulatory support (MCS) at risk of complications after MCS. The INTERMACS scale goes from 1-7, where INTERMACS 1 is "crash and burn" and 7 is stable at home with some symptoms.
  Participants
    1 | 3 | 1 | 1 | 0 | 5
    2 | 6 | 5 | 0 | 0 | 11
    3 | 3 | 2 | 0 | 0 | 5
    4 | 0 | 0 | 0 | 0 | 0
    5 | 0 | 0 | 0 | 0 | 0
    6 | 0 | 1 | 0 | 0 | 1
    Unknown | 0 | 1 | 0 | 0 | 1
LVAD Type [Count of Participants; unit: Participants]
  HeartMate II | 0 | 0 | 1 | 0 | 1
  Heartware Ventricular Assisted Device (HVAD) | 3 | 5 | 0 | 0 | 8
  Heart Mate III | 9 | 5 | 0 | 0 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Markers of Angiogenesis - Angiopoietin 1/2 and VEGF
Description: Markers of angiogenesis and inflammation will be measured on customized Luminex assay panels. These will include Angiopoietin-1 (ng/mL), Angiopoietin-2 (ng/mL), and VEGF (ng/mL).
Time Frame: Markers will be measured at baseline at randomization, and at 3 months, 6 months, and 12 months after randomization.
Population: as for baseline characteristics
Arm/Group | Primary Prevention Intervention | Primary Prevention Non-Intervention | Secondary Prevention Intervention | Secondary Prevention Non-Intervention
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Change in Markers of Angiogenesis - TNF-alpha
Description: Markers of angiogenesis and inflammation will be measured on customized Luminex assay panels. These will include TNF-alpha (pg/mL).
Time Frame: Markers will be measured at baseline at randomization, and at 3 months, 6 months, and 12 months after randomization.
Population: as for baseline characteristics
Arm/Group | Primary Prevention Intervention | Primary Prevention Non-Intervention | Secondary Prevention Intervention | Secondary Prevention Non-Intervention
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Change in Markers of Inflammation - C-Reactive Protein
Description: Markers of angiogenesis and inflammation will be measured on customized Luminex assay panels. These will include c-reactive protein (mg/dL).
Time Frame: Markers will be measured at baseline at randomization, and at 3 months, 6 months, and 12 months after randomization.
Population: as for baseline characteristics
Arm/Group | Primary Prevention Intervention | Primary Prevention Non-Intervention | Secondary Prevention Intervention | Secondary Prevention Non-Intervention
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Rates of Gastrointestinal Bleeding
Description: Rates of Gastrointestinal Bleeding will be assessed.
Time Frame: Rates of bleeding will be measured at 3 months, 6 months, and 12 months after randomization.
Population: Study terminated by PI for low/no enrollment. All efforts were taken to gather all possible data.
Arm/Group | Primary Prevention Intervention | Primary Prevention Non-Intervention | Secondary Prevention Intervention | Secondary Prevention Non-Intervention
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Changes in the Microbiome
Description: The microbiome will be assessed using rectal swabs. The swabs will be analyzed to determine the bacterial species present at each time point.
Time Frame: The microbiome will be assessed at baseline at randomization, and at 3 months, 6 months, and 12 months after randomization.
Population: as for baseline characteristics
Arm/Group | Primary Prevention Intervention | Primary Prevention Non-Intervention | Secondary Prevention Intervention | Secondary Prevention Non-Intervention
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected within the first year of the study.
Description: Patients were assessed at clinic for medication compliance and self-reported medication side effects, in addition to follow-up calls for any additional medication side effects.
  Study terminated by PI for low/no enrollment. All efforts were taken to gather all possible data.
Arm/Group | Primary Prevention Intervention | Primary Prevention Non-Intervention | Secondary Prevention Intervention | Secondary Prevention Non-Intervention
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/10 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Prevention Intervention (N=12) | Primary Prevention Non-Intervention (N=10) | Secondary Prevention Intervention (N=1) | Secondary Prevention Non-Intervention (N=0)
nausea and indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated by PI for low/no enrollment prior to primary and secondary endpoints. All efforts were taken to gather all possible data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT03784963/Prot_SAP_000.pdf